CLINICAL TRIAL: NCT04376125
Title: Suboccipital Inhibition in Tension Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de León (Other)
Collaborators: Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Cristina Blanco Ortega, principal investigator, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71441538L
Record Dates: First submitted 2019-02-24; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Tension Headache
Keywords: tension headache; suboccipital inhibition
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital inhibition in tension headache (Experimental): Two groups of patients suffering from tension headache associated with cervicalgia are selected.
  The control group performs conventional therapy. The experimental group performs conventional therapy plus the technique of suboccipital inhibition
  Interventions: Other: Suboccipital inhibition in tension headache
- study of results (Active Comparator): We compared data from both groups
  Interventions: Other: Suboccipital inhibition in tension headache

INTERVENTIONS:
Other: Suboccipital inhibition in tension headache — Deep maneuver of myofascial induction in the suboccipital muscles

SUMMARY:
The researchers will carry out a randomized experimental study. Participants in the experimental group will receive a treatment based on suboccipital inhibition technique in addition to conventional treatment. Participants in the control group will only receive the conventional treatment. The existence of significant differences in both groups will be analyzed.

DETAILED DESCRIPTION:
Conventional therapy will consist of microwaves, interference currents, and manual therapy.

ELIGIBILITY:
Inclusion Criteria:

* pathology tension headache associated with cervicalgia

Exclusion Criteria:

* pathology of nervous system

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale for Pain | immediately before starting the intervention and after the last session of the intervention, that is, 2 weeks from the start
  a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst imaginable pain" (score of 10)

SECONDARY OUTCOMES:
Change in Six-item Headache Impact Text | immediately before starting the intervention and after the last session of the intervention, that is, 2 weeks from the start
  A global measure of adverse headache impact. The final HIT-6 score is obtained from simple summation of the six items and ranges between 36 and 78, with larger scores reflecting greater impact.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Blanco Ortega, physiotherap, Principal Investigator — Universidad de León
Locations (1):
- Cristina Blanco Ortega, León, Spain

IPD SHARING:
Plan to Share IPD: No